CLINICAL TRIAL: NCT00313859
Title: Phase II Study of Simvastatin Plus Irinotecan, Fluorouracil, and Leucovorin(FOLFIRI) for Metastatic Colorectal Cancer
Brief Title: Phase II Study of Simvastatin Plus Irinotecan, Fluorouracil, and Leucovorin(FOLFIRI) for Metastatic CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2005-08-011
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer; Metastasis
Keywords: colorectal cancer; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Simvastatin

INTERVENTIONS:
Drug: simvastatin

SUMMARY:
This trial is designed to assess the tolerability and efficacy of simvastatin plus FOLFIRI (irinotecan, 5-FU, leucovorin) in metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
Progress in treatment for metastatic CRC has undoubtedly been achieved in the past decade. Until 1985, 5-fluorouracil (5-FU) was the only agent available for the treatment of metastatic CRC. Several trials have attempted to enhance the activity of bolus 5-FU, by the addition of levamisole or interferon. Despite of these attempts, no survival advantage was established until the introduction of the newer cytotoxic drugs. The addition of folinic acid (FA) to 5-FU, the use of infusional rather than bolus 5-FU, and the combination of new active agents such as irinotecan and oxaliplatin with 5-FU/FA have resulted in an increase in activity of 5-FU. In trials of current combination regimens as first-line therapy, response rates exceeding 30% and median survival duration longer than 16 months have been reported. In all, despite of rapid advances in the treatment of metastatic CRC during the last decade, the efficacy of treatment still needs to be improved. One potential way of increasing the survival of metastatic CRC patients is the introduction of a novel targeting agent to the standard cytotoxic regimen such as IFL (irinotecan, fluorouracil, and leucovorin). An increasingly recognized molecular target for anticancer treatment is the rate-limiting enzyme of the mevalonate pathway, 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase. The end products of the mevalonate pathway are required for a number of essential cellular functions such as sterols for membrane integrity, ubiquinone for cell respiration, geranylgeranyl isoprenoids for covalent bindings to the ras family, dolichol for glycoprotein synthesis, and isopentenyladenine for tRNA function and protein synthesis. Fortunately, inhibitors of the key enzyme, the statins, are well established and have been used safely in the clinic for the treatment of hypercholesterolemia for decades. Therefore, HMG-CoA reductase may be a decent molecular target for anti-cancer therapy and statins may be readily applicable to the clinic once its potential role as an anticancer drug is established. The statins have recently gained attractions from medical oncologists because large retrospective analyses for efficacy trials of statins in coronary artery disease have shown that not only are these agents able to reduce cardiac disease-related mortality, but cancer incidence is also reduced by 28 - 33 %.

In all, further clinical trials investigating on combining the standard treatment with these novel molecular targeting agents, the statins, are definitely warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic colorectal cancer
2. Age ≥ 18
3. ECOG performance status 0 - 2
4. At least one measurable lesion
5. Minimum life expectancy of 12 weeks
6. Adequate bone marrow reservoir (ANC ≥ 1500/㎕, platelet ≥ 100,000/㎕)
7. Adequate renal function (serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 50 min/ml)
8. Adequate liver functions (serum bilirubin ≤ 1.5 mg/dl, AST/ALT ≤ 3 times upper normal limits)
9. No prior lipid-lowering therapy with statins less than 1 year before study entry
10. No prior chemo- or immunotherapy for metastatic CRC (adjuvant chemotherapy or chemoradiation therapy more than 6 months before study entry is permitted)
11. Written informed consent

Exclusion Criteria:

1. Active infection requiring antibiotics therapy
2. Pregnancy and/or lactation
3. Other serious illness or medical condition not appropriate for chemotherapy, especially cardiovascular disease
4. Metastatic brain lesions
5. Receipt of radiotherapy within 2 weeks before the initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
overall response rate

SECONDARY OUTCOMES:
progression-free survival
overall survival
toxicity
duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea